CLINICAL TRIAL: NCT03065257
Title: Endoscopic Resection: A Retrospective and Prospective Multicenter Registry
Brief Title: Endoscopic Resection Multicenter Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Michel Kahaleh, Chief of Endoscopy, Weill Medical College of Cornell University
Other Study IDs: 1701017930
Record Dates: First submitted 2017-02-16; First posted 2017-02-27 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Gastrointestinal Neoplasms; Gastrointestinal Disease; Gastric Cancer; Gastric Neoplasm; Gastric Polyp; Esophageal Neoplasms; Duodenal Neoplasms; Duodenal Polyp; Stomach Neoplasm; Stomach Polyp; Neoplasms; Colon Polyp; Colon Neoplasm
Keywords: EMR; ESD; Resection; STER; EFTR; Submucosal dissection; Endoscopic resection
MeSH Terms: conditions — Gastrointestinal Neoplasms; Gastrointestinal Diseases; Stomach Neoplasms; Polyposis, Gastric; Esophageal Neoplasms; Duodenal Neoplasms; Neoplasms; Colonic Polyps; Colonic Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopic Resection: Patients undergoing Endoscopic Resection
  Interventions: Procedure: Endoscopic Resection

INTERVENTIONS:
Procedure: Endoscopic Resection — Any Endoscopic resection for Gastrointestinal disorders including neoplasms.

SUMMARY:
This is a retrospective and prospective multicenter registry to collect long-term data (1 year) on patients who have or will undergo Endoscopic resection such as EMR, ESD, EFTR, STER, etc. within the gastrointestinal tract for endoscopic treatment of early gastrointestinal neoplasms involving the resection of the superficial layers, mucosa and submucosa, of the tract wall.

Subjects will be consented for medical chart review.

The purpose of this retrospective and prospective registry is to assess long term data on efficacy, safety and clinical outcome of Endoscopic Resection within the gastrointestinal tract (1 year).

The registry will evaluate efficacy, technical feasibility, clinical outcome, safety profile and overall clinical management through medical chart review. The procedures the investigators are evaluating are all clinically indicated and will not be prescribed to someone to participate in this registry study.

DETAILED DESCRIPTION:
Endoscopic resection can be an appropriate approach in early neoplasms, challenging adenomas or sub-epithelial lesions. Endoscopic resection can be considered as a less invasive approach than surgery. Moreover, endoscopic resection can be available to patients who are ineligible for surgery or who have refused more aggressive surgical intervention.

The study investigators would collect data on a large sample size of subjects undergoing various endoscopic resection procedures such as EMR (Endoscopic Mucosal Resection), ESD (Endoscopic submucosal dissection), STER (Submucosal tunneling endoscopic resection, and EFTR (Endoscopic full-thickness resection). Clinical metrics will be recorded including procedure times, length of follow-up, specific tumor characteristics, resection method, pathology results, procedural complications, additional therapy required, and disease-free survival time.

Currently, there is limited multi-center data on endoscopic resection outcomes in western populations.

Evaluation of these measurement would help the investigators compare them to conventional treatment modalities within current tertiary facilities; and consequently help the investigators identify appropriate treatment techniques and improve clinical management of patients at WCMC-NYPH.

The purpose of this retrospective and prospective registry is to assess long term data on efficacy, safety and clinical outcome of Endoscopic Resection within the gastrointestinal tract (1 year).

ELIGIBILITY:
Inclusion Criteria:

* Any patient who is considering undergoing endoscopic resection within 6 months, or has undergone clinically indicated endoscopic resection within the past 6 months
* Above or equal to 18 years of age.

Exclusion Criteria:

* Any patient who has not undergone or will undergo endoscopic resection
* Below 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing Endoscopic resection procedures as part of their clinically indicated care
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-03-15 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with reduction in clinical symptoms | 6 months from procedure
  To assess resolution of symptoms of all Endoscopic resection procedures at 6 months

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 30 days post procedure
  Number of subjects with Adverse Events; Type, frequency and intensity of adverse events within 30 days of procedure

OTHER OUTCOMES:
Number of participants with successful completion of treatment | 30 days post procedure
  Number of participants with successful completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michel Kahaleh, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No IPD Sharing